CLINICAL TRIAL: NCT03297489
Title: A Pilot Study of Feasibility of Performing Intravital Microscopy in Patients With Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Intravital Microscopy in Evaluating Patients With Primary Peritoneal, Fallopian Tube, or Stage IA-IV Ovarian Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 43717; NCI-2017-01459 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 43717 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Stage I Ovarian Cancer; Stage IA Ovarian Cancer; Stage IB Ovarian Cancer; Stage IC Ovarian Cancer; Stage II Ovarian Cancer; Stage IIA Ovarian Cancer; Stage IIB Ovarian Cancer; Stage IIC Ovarian Cancer; Stage III Ovarian Cancer; Stage IIIA Ovarian Cancer; Stage IIIB Ovarian Cancer; Stage IIIC Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Fluorescein; Fluoresceins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (intravital microscopy) (Experimental): Patients receive fluorescein sodium injection IV. Patients also undergo observation of primary and metastatic tumors via microscopy over 15-20 minutes during the course of standard of care surgery.
  Interventions: Procedure: Diagnostic Microscopy; Drug: Fluorescein Sodium Injection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Diagnostic Microscopy — Undergo observation via intravital microscopy
Drug: Fluorescein Sodium Injection — Given IV
  Other Names: AK-Fluor; Fluorescite
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well intravital microscopy works in evaluating patients with primary peritoneal, fallopian tube, or stage IA-IV ovarian cancer. Intravital microscopic evaluation of tumor blood vessels, blood flow, immune cell interactions, and drug uptake may be eventually visualized and may lead to valuable prognostic information.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of performing intravital microscopy on accessible human ovarian, primary peritoneal and fallopian tube cancers during their standard course of treatment (i.e., surgical debulking).

SECONDARY OBJECTIVES:

I. To determine the blood flow velocity of the tumor vessels and tissue penetration of fluorescein as a marker of tumor vessel permeability.

OUTLINE:

Patients receive fluorescein sodium injection intravenously (IV). Patients also undergo observation of primary and metastatic tumors via microscopy over 15-20 minutes during the course of standard of care surgery.

After completion of study, patients are followed up for 30 days, at 1-3 weeks, and then up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Suspicion of gynecological malignancy that requires a standard of care surgical resection in the operating room;
* Have measurable lesion in the pelvis or abdomen, at a minimum of 0.5 cm in diameter on standard of care pre operative imaging studies (CT, MRI or PET scan),
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Serum Creatinine <= 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN (using Cockcroft-Gault Equation), GFR can also be used in place of creatinine or CrCl.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any known allergy or prior reaction to fluorescein
* Nursing female subjects
* Liver dysfunction; normal liver function defined as total bilirubin within normal institutional limits and aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to undergo observational study (may also include preoperative testing results including electrocardiography (EKG), chest x-ray, or pulmonary function tests that preclude a wide excision in the operating room)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Fluorescein within the tumor vessels | Up to 2 years
  Will visualize fluorescein within the tumor vessels.
Identification of tumor vessels | Up to 2 years
  Will identify tumor vessels.
Tumor vessel diameter | Up to 2 years
  Will measure tumor vessel diameters.
Vessel density | Up to 2 years
  Will determine vessel density per 10 x field.

SECONDARY OUTCOMES:
Blood flow velocity of the tumor vessels | Up to 2 years
  Will assess the ability to measure the blood flow velocity of the tumor vessels.
Tissue penetration of fluorescein | Up to 2 years
  Will measure tissue penetration of fluorescein as a marker of tumor vessel permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States